CLINICAL TRIAL: NCT04733469
Title: EMPOWER 3: Improving Palliative Care Health Literacy and Utilization
Acronym: EMPOWER 3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: American Cancer Society, Inc. (Other); University Medical Center-New Orleans (Unknown)
Responsible Party: Principal Investigator, Michael Hoerger, PhD, MSCR, Associate Professor of Psychology, Psychiatry, and Oncology, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 134579-RSG-20-058-01-PCSM
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia Psychoeducational Intervention + Enhanced Usual Care (Experimental): Intervention participants receive the Multimedia Psychoeducational Intervention in addition to Enhanced Usual Care
  Interventions: Behavioral: Multimedia Psychoeducational Intervention; Behavioral: Enhanced Usual Care
- Enhanced Usual Care (Other): Control participants receive Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Multimedia Psychoeducational Intervention — The Multimedia Psychoeducational Intervention includes a multimedia educational video plus additional resources to reinforce the video content. The Multimedia Psychoeducational Intervention includes the following:
  * A multimedia educational video about palliative care that is individually tailored to each patient's level of education and health literacy
  * Take-home and online copies of the video for repeat viewing
  * A video summary
  * A question prompt list patients can use to ask clinicians more questions about palliative care
  * Contact information and brochures for local palliative care programs
  Arms: Multimedia Psychoeducational Intervention + Enhanced Usual Care
Behavioral: Enhanced Usual Care — Enhanced Usual Care refers to usual care plus minor enhancement to improve quality and standardization. Enhanced Usual Care includes the following:
  * Usual care
  * A packet of flyers and handouts with general information on psychosocial oncology services derived from the American Society of Clinical Oncology (ASCO), Center to Advance Palliative Care (CAPC), and American Cancer Society (ACS)

SUMMARY:
Through this award, Michael Hoerger, PhD, MSCR, a psychologist at the Tulane Cancer Center in Louisiana, will lead a study called EMPOWER 3 designed to test an educational intervention to help patients understand palliative care, use it, and feel better emotionally and physically. Participants will be adults with serious cancer diagnoses. Participants will be randomized into two groups. Patients in the control group will get enhanced usual care, meaning standard cancer care and several additional healthcare-related brochures. Patients in the intervention group will get enhanced usual care plus an educational video developed by the investigators and other materials designed to increase understanding and use of palliative care. Family members of patients in the intervention group may also attend if desired. The investigators will track participants' understanding of palliative care, attitudes toward palliative care, symptoms over 6 months of follow-up, and palliative care utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age 18 or older
2. Meets criteria for 2a or 2b. 2a) The patient's doctor believes they may be appropriate for palliative cancer care OR 2b) The patient has a new diagnosis, recurrence, or progression of cancer in the past 90 days AND any of the following:

   * Advanced cancer, such as:

     * Lung Cancer: Stage IIIB or IV non-small cell, or extensive stage small cell
     * Breast Cancer: Stage IV
     * Gastrointestinal (GI) Cancers: Unresectable stage III or stage IV
     * Genitourinary (GU) Cancers: Stage IV
     * Melanoma: Stage IV
     * Hematologic Malignancies

       * Leukemia (e.g., acute myeloid leukemia [AML], acute lymphoblastic leukemia [ALL], chronic myeloid leukemia (CML), chronic lymphocytic leukemia [CLL]): advanced stage, treatment refractory, poor prognosis cell type or chromosomal abnormalities, older age
       * Lymphoma: Stage IV or treatment refractory Hodgkin's disease or non-Hodgkin's lymphoma Multiple Myeloma: elevated β2-microglobulin, albumin <3.5, PCLI >1%, CRP >6µg/mL, elevated LDH, plasmablastic morphology, or abnormal chromosome 13
   * Advanced heart, lung, renal (kidney), or liver disease
   * Two or more severe symptoms (≥7 on 0-10 scale): pain, tiredness, drowsiness, nausea, bad appetite, shortness of breath, depression, or anxiety
3. Patient can understand spoken or written English
4. Patient receives care in southeast Louisiana

Exclusion Criteria:

* Known history of receiving specialty palliative care or hospice
* Significant psychiatric or other co-morbid disease that would prohibit informed consent or participation in the study
* Unlikely to complete any follow-up surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Palliative Care Knowledge Scale (PaCKS) | Post-test of Visit 1, typically day 1
  Percentage correct on 13 items; higher scores indicate greater knowledge

SECONDARY OUTCOMES:
Aim 2a: Palliative Care Attitudes Scale (PCAS-9) | Post-test of Visit 1, typically day 1
  Total score from 0-36; higher scores indicate more positive attitudes
Aim 2b: Palliative Care Utilization | Up to 90 days
  Utilization of palliative care (presence/absence)
Aim 3a: Patient-Reported Outcome Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions | Follow-up at 14, 90, and 180 days
  Total score from 8-40 on 8 items from PROMIS self-efficacy for managing symptoms and self-efficacy for managing emotions items banks; higher scores indicate greater self-efficacy
Aim 3b: PROMIS Emotional Distress | Follow-up at 14, 90, and 180 days
  Total score from 8-40 on 8 items from the PROMIS Depression and Anxiety item banks; higher scores indicate greater symptom severity
Aim 3c: Edmonton Symptom Assessment Scale (ESAS)-Physical | Follow-up at 14, 90, and 180 days
  Total score from 0-60 on 6 ESAS ratings of pain, tiredness, drowsiness, nausea, poor appetite, and difficulty breathing; higher scores indicate greater symptom severity

OTHER OUTCOMES:
Exploratory: Brief COPE Inventory | Follow-up at 14 days
  Total score from 6-24 on 6 Brief COPE Inventory items measuring denial, acceptance (reverse-coded), and self-blame; higher scores indicate less effective coping
Exploratory: PROMIS Anger | Follow-up at 90 days
  Total score from 2-10 on 2 items from the PROMIS Anger item bank; higher scores indicate more anger
Exploratory: PROMIS Positive Affect | Follow-up at 90 days
  Total score from 2-10 on 2 items from the PROMIS Positive Affect item bank; higher scores indicate more positive affect
Exploratory: PROMIS Stress | Follow-up at 90 days
  Total score from 4-20 on 4 items from the PROMIS Stress item bank; higher scores indicate more stress
Exploratory: PROMIS General Self-Efficacy | Follow-up at 90 days
  Total score from 4-20 on 4 items from the PROMIS General Self-Efficacy item bank; higher scores indicate more stress
Exploratory: Medication Adherence | Follow-up at 90 days
  Rating from 1-6 (Very poor to Excellent) for quality of medication adherence in the past 30 days; higher scores indicate better adherence
Exploratory: PROMIS Emotional Support | Follow-up at 180 days
  Total score from 2-10 on 2 items from the PROMIS Emotional Support item bank; higher scores indicate more emotional support
Exploratory: PROMIS Cognitive Function | Follow-up at 180 days
  Total score from 4-20 on 4 items from the PROMIS Cognitive Function item bank; higher scores indicate better cognitive function
Exploratory: PROMIS Meaning and Purpose | Follow-up at 180 days
  Total score from 2-10 on 2 items from the PROMIS Meaning and Purpose item bank; higher scores indicate more meaning and purpose
Exploratory: Quality of Life in Neurologic Disorders (Neuro-QoL) Concern with Death and Dying | Follow-up at 180 days
  Total score from 2-10 on 2 items from the Neuro-QoL Concern with Death and Dying item bank; ; higher scores indicate more concern

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoerger, PhD, MSCR, MBA, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - University Medical Center, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared with other researchers upon completing a data usage agreement signed by all participating universities.
Supporting Information: Study Protocol, ICF
Time Frame: By the study end date, available for at least 3 years.
Access Criteria: Contact the Study PI